CLINICAL TRIAL: NCT06432205
Title: The Effect of Multi-Disciplinary Team Plus Shared-Decision Making on Survival Benefit of Advanced Gastric Cancer - a Single Center, Non-randomized, Prospective, Controlled Study
Brief Title: The Effect of MDT Plus SDM on Survival Benefit of Advanced Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023YJZ66
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer
Keywords: multi-disciplinary Team; shared-decision making; surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgery group: metastatic gastric cancer patients who are assessed as having the opportunity for surgery finally choose to undergo surgery after MDT plus SDM.
  Interventions: Procedure: surgery
- non-surgery group: metastatic gastric cancer patients who are assessed as having the opportunity for surgery finally choose not to undergo surgery after MDT plus SDM.

INTERVENTIONS:
Procedure: surgery — any forms of surgery, such as all tumor resection, partial tumor resection and palliative tumor resection surgery
  Groups: surgery group

SUMMARY:
The goal of this observational study is to learn about the long-term effect of surgery in metastatic gastric cancer patients who are accessed as having opportunity for surgery under Multi-disciplinary Team (MDT) evaluation. The main question it aims to answer is:

Does surgery extend survival time in metastatic gastric cancer patients who are accessed as having opportunity for surgery under Multi-disciplinary Team (MDT) evaluation?

DETAILED DESCRIPTION:
Select metastatic gastric cancer patients that have the opportunity to undergo any forms of surgery through MDT. Then further evaluate these patients' risks and benefits. Let patients make their finally decision through shared-decision making (SDM). According to the actual decision, the patients are divided into surgery group and non-surgery group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Participate in the formal MDT discussion and evaluate feasible surgical treatment;
* Gastric adenocarcinoma or gastroesophageal junction adenocarcinoma confirmed by histology;
* Immunotherapy must be received during the treatment;
* At least 1 distant metastatic organs, and the number of metastases is ≥1;
* The subject line blood routine (within 7 days) and biochemical indicators (within 14 days) meet the following standards:

hemoglobin≥90g/L； absolute count of neutral granulocytes (ANC) ≥1.5×10^9/L； platelets≥100×10^9/L； Alt, AST≤ 2.5 times the normal upper limit，≤5 times the normal upper limit value (with liver metastasis)； ALP ≤ 2.5 times the normal upper limit，≤5 times the normal upper limit (with liver or bone metastasis)； total bilirubin<1.5 times the normal upper limit value of serum； serum creatinine<1.5 times normal upper limit； albumin≥30g/L；

* ECOG 0 ～ 1 point;
* The expected life span is ≥3 months;
* Cardiopulmonary function is basically normal;
* Women and spouses of childbearing age are willing to adopt effective contraceptive methods.

Exclusion Criteria:

* Those who do not meet the above selected standards or have chemotherapy contraindications;
* Combined with other primary malignant tumors;
* Pregnancy, lactating women or women of childbearing age and spouses refuse to adopt effective contraceptive methods;
* History of organ transplantation (including bone marrow autologous transplantation and peripheral stem cell transplantation);
* History of long -term treatment of steroids (Note: Short -term users discontinue drugs> 2 weeks can be selected);
* History of peripheral nervous system disorders or obvious mental disorders and central nervous system disorders;
* Accompanied by severe infection;
* Accompanied by swallowing difficulties, complete or incomplete digestive tract obstruction, gastrointestinal bleeding, perforation, etc.;
* Severe liver disease (such as liver cirrhosis, etc.), kidney disease, respiratory disease, or chronic system diseases such as diabetes, hypertension, high blood pressure;
* Coronary heart disease with obvious clinical symptoms, such as: congestive heart failure, obvious symptoms, cardiac disorders, hypertension, or myocardial infarction seizures, or inadequate heart function within 6 months;
* Persons without legal capacity, medical or ethical reasons affecting the continuation of research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient in Beijing Cancer Hospital
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
overall survival | From diagnosis of metastatic gastric cancer to any cause of death，assessed up to 5 years

SECONDARY OUTCOMES:
progression free survival | From diagnosis of metastatic gastric cancer to tumor progression or any cause of death, assessed up to 2 years
safety of surgery | after surgery, assessed up to 24 weeks
  any grade of adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China